CLINICAL TRIAL: NCT07105215
Title: A Multicenter Phase I/II Clinical Study to Evaluate the Safety and Efficacy of RC278 for Injection in the Treatment of Locally Advanced Unresectable or Metastatic Malignant Solid Tumor
Brief Title: A I/II Phase Clinical Study to Evaluate the Safety and Efficacy of RC278 in the Treatment of Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC278-C001
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RC278 (Phase I, dose escalation) (Experimental): There are five escalating dose cohorts.
  Interventions: Drug: RC278
- RC278 (Phase I, dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored.
  Interventions: Drug: RC278
- RC278 (Phase I, dose optimization) (Experimental): Based on the safety, pharmacokinetic (PK), and efficacy data from the subjects, select at least two dose levels and randomly assign subjects in a 1:1 ratio to determine the recommended Phase II dose (RP2D) for entering the Phase II stage.
  Interventions: Drug: RC278
- RC278 (Phase II) (Experimental): In the multi-indication cohort expansion phase, further assess the efficacy and safety of RC278 in various cancer types using the RP2D.
  Interventions: Drug: RC278

INTERVENTIONS:
Drug: RC278 — Intravenous (IV) administration of RC278 Q3W. Patients will continue treatment until unacceptable toxicities, disease progression, or any criterion for withdrawl from the study.
  Other Names: RC278 For Injection

SUMMARY:
The primary objective is to evaluate the safety and tolerability of RC278; determine the maximum tolerated dose (MTD) and/or maximum administered dose (MAD) of RC278; and determine the recommended phase 2 dose (RP2D)， and assess the efficacy of RC278 at the RP2D dose;

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, sign the informed consent form, and be able to adhere to the study protocol;
2. Age between 18 and 75 years (including 18 and 75 years);
3. ECOG PS score of 0 or 1;
4. Expected survival ≥12 weeks;
5. According to RECIST v1.1 criteria, based on imaging examinations, there is at least one measurable target lesion;
6. Sufficient bone marrow, liver, kidney, and blood clotting function

Exclusion Criteria:

1. Pregnant, breastfeeding, or intending to become pregnant subjects.
2. Subjects with brain metastases.
3. Subjects with unresolved toxicities from prior anti-tumor therapy not recovered to NCI-CTCAE v5.0 Grade 1.
4. Subjects with known hypersensitivity or delayed allergic reactions to any component of the investigational drug or similar drugs.
5. Subjects with acute, chronic, or symptomatic infections.
6. Subjects with uncontrolled cardiovascular diseases.
7. Subjects with confirmed or suspected interstitial lung disease (ILD), drug-related pneumonia, radiation pneumonitis, severely impaired pulmonary function, or other pulmonary diseases.
8. Subjects with a history of cirrhosis (Child-Pugh B or C class).
9. Subjects with active inflammatory bowel disease.
10. Subjects with uncontrolled diabetes (HbA1c ≥ 10%).
11. Subjects who experienced arterial/venous thromboembolic events, deep vein thrombosis, pulmonary embolism, or stroke within 6 months prior to the first dose.
12. Subjects with pericardial effusion or cardiac tamponade, or third-space fluid accumulation, which, in the investigator's judgment, cannot be controlled or stabilized by drainage or other methods.
13. Subjects with active autoimmune diseases requiring systemic treatment within the past 2 years.
14. Subjects with a history of other invasive malignancies within 5 years prior to the first dose, or evidence of residual disease from a previously diagnosed malignancy.
15. Subjects with a history of other acquired or congenital immunodeficiency diseases or organ transplantation.
16. Subjects with a history or current diagnosis of uncontrolled psychiatric disorders.
17. Subjects with poor adherence, who are unlikely to comply with the trial procedures.
18. Subjects with any other diseases, metabolic abnormalities, physical examination abnormalities, or laboratory abnormalities, which, in the investigator's judgment, raise suspicion of an underlying condition making the subject unsuitable for the investigational drug, or which may affect the interpretation of the study results, or place the subject at high risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 24 months
  DLT is defined as the adverse events (AEs) occurring during the DLT observation period that the investigator determines to be related to the RC278 treatment.
Incidence and severity of adverse events/serious adverse events (graded according to NCI CTCAE v5.0) | 24 months
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the CTCAE Version 5.0].
Determine RP2D of RC278 | 24 months
  To determine the RP2D for further evaluation of RC278 in subjects with advanced solid tumor.
MTD and/or MAD | 24 months
  To determine the MTD and/or MAD for further evaluation of RC278 in subjects with advanced solid tumor.
Investigator assessed ORR according to RECIST v1.1 criteria | 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institute, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Luoyan, Henan
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, China, Wuhan, Hu'Nan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, China, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Tumor Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School Of Medicine, Hangzhou
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Jinan Central Hospital, Jinan
  - Shanxi Cancer Hospital, Taiyuan
  - Henan Cancer Hospital, Zhengzhou